CLINICAL TRIAL: NCT00003723
Title: Phase II Study of Gemcitabine and Cisplatin in Unresectable Malignant Mesothelioma
Brief Title: S9810: Gemcitabine Plus Cisplatin in Treating Patients With Malignant Mesothelioma of the Pleura That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066832; SWOG-S9810 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-06-24 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Malignant Mesothelioma
Keywords: advanced malignant mesothelioma; epithelial mesothelioma; sarcomatous mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Solitary Fibrous Tumor, Pleural | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine/Cisplatin (Experimental): Gemcitabine 1000 mg/m^2 days 1, 8 15 (q 28 days) cisplatin 30 mg/m^2 days 1, 8, 15 (q 28 days)
  Interventions: Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Gemcitabine 1000 mg/m^2 days 1, 8 15 (q 28 days)

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of gemcitabine plus cisplatin in treating patients with malignant mesothelioma of the pleura that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate overall survival and confirmed and unconfirmed complete and partial response in patients with unresectable malignant mesothelioma of the pleura treated with gemcitabine plus cisplatin. II. Evaluate the qualitative and quantitative toxicities of this regimen in this patient population.

OUTLINE: Patients receive gemcitabine IV over 30 minutes, immediately followed by cisplatin IV over 30 minutes on days 1, 8, and 15. Courses are repeated every 28 days. Treatment continues in the absence of unacceptable toxicity or disease progression. Patients with a complete response receive 2 additional courses of therapy. Patients are followed every 6 months until death.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study within 25 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed diagnosis of unresectable malignant mesothelioma of the pleura Epithelial, fibrosarcomatous, or mixed type Bidimensionally measurable disease No CNS metastases

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: SWOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Platelet count at least lower limit of normal Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT or SGPT no greater than 2.5 times upper limit of normal (ULN) Renal: Creatinine no greater than 2 times ULN AND Creatinine clearance at least 60 mL/min Other: Not pregnant or nursing Fertile patients must use effective contraception No other prior malignancy within the past 5 years except adequately treated basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or adequately treated stage I or II cancer currently in complete remission Must have chest x-ray within the past 28 days

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy No other concurrent chemotherapy Endocrine therapy: Concurrent hormones for non-disease-related conditions allowed Concurrent steroids for antiemesis, adrenal failure, or septic shock allowed Radiotherapy: No prior radiotherapy No concurrent radiotherapy Surgery: At least 4 weeks since prior major surgery and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 1999-02; Primary Completion 2007-06 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Estimate overall survival | monthly while patient on treatment. Once off treatment every 6 months

SECONDARY OUTCOMES:
qualitative and quantitative toxicities | week 1, 2, 3 (q 28 days)
confirmed and unconfirmed complete and partial response | every 8 weeks until progression

CONTACTS AND LOCATIONS:
Overall Officials: Robert N. Taub, MD, PhD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (84):
- United States (84):
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - University of California Davis Medical Center, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- [Result] Kalmadi SR, Rankin C, Kraut MJ, Jacobs AD, Petrylak DP, Adelstein DJ, Keohan ML, Taub RN, Borden EC. Gemcitabine and cisplatin in unresectable malignant mesothelioma of the pleura: a phase II study of the Southwest Oncology Group (SWOG 9810). Lung Cancer. 2008 May;60(2):259-63. doi: 10.1016/j.lungcan.2007.09.018. Epub 2007 Nov 19. PMID 18006112